CLINICAL TRIAL: NCT04028414
Title: Effects of Early Weight Bearing on Rehabilitation Outcomes in Patients With Traumatic Ankle and Tibial Plateau Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-18-1-0810
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Weight Bearing (Experimental): Patients with ankle fractures will be instructed to weight bear as tolerated (WBAT) while in a boot with a heel to toe normal gait and wean from walker or crutches to a cane or no support device. At the 6 week post op visit, patients with ankle fractures will be instructed to wean from the boot and continue full weight bearing as tolerated until full weight bearing is achieved. Patients with plateau fractures will be instructed to begin WBAT until full weight bearing is achieved.
  Interventions: Other: Early Weight Bearing
- Delayed Weight Bearing (No Intervention): Patients with ankle fractures will be instructed to touch-down (toe touch or foot flat) weight bear (approximately 10% of body weight) while in the boot for. Patients will be instructed to keep foot off of floor or set ball of foot or heal on ground for balance using walker or crutches at all times. After the 6 week post op visit, patients may begin weight bearing as tolerated. Patients with tibial plateau fractures will be instructed to touch down (toe touch or foot flat) weight bear (approximately 10% of body weight) for at least 6 weeks. After the 6 week post op visit, patients may begin weight bearing as tolerated until full weight bearing is achieved.

INTERVENTIONS:
Other: Early Weight Bearing — Patients will be instruction to weight bear as tolerated while in a boot.
  Arms: Early Weight Bearing

SUMMARY:
The overall objective of this study is to compare outcomes following early versus delayed weight bearing for adult patients operatively treated for an ankle fracture without syndesmotic fixation. Additionally, early weight bearing will be tested in patients with unicondylar plateau fractures that do not involve joint impaction in the context of a pilot study.

DETAILED DESCRIPTION:
The purpose of this multi-center, randomized controlled trial (RCT) is to compare outcomes following early versus delayed weight bearing among individuals with a traumatic ankle fracture. This study will enroll patients ages 18 or older surgically treated for an ankle fracture or fracture dislocation (without syndesmosis) at participating civilian trauma centers and military treatment facilities. Eligible patients will be identified during hospitalization for definitive treatment and enrolled prior to discharge or at the first post op clinic visit. Patients that consent to participate will complete a baseline assessment at the first post op clinic visit and will be randomized to early versus delayed weight bearing. Both treatment groups will receive standardized exercises that can be done at home or with a therapist. Outcomes will be evaluated at 6 weeks, 3, 6 and 12 months following definitive fracture fixation. All 6 week, 3 and 6 month evaluations will take place in the surgeon's outpatient clinic and involve clinical and radiographic assessments of healing as well as functional outcome surveys. The 12 month evaluation will be conducted by phone except for individuals who were judged not to be healed (clinically or radiographically) at 6 months; these participants will be asked to return for their 12 month evaluation (to assess healing). Simultaneously, a pilot RCT will be conducted in patients 18 or older surgically treated with a unicondylar plateau fracture without joint impaction.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 or older
2. Surgically treated open or closed fractures of the ankle (OTA Codes 44A,B,C) meeting one of the following criteria:

   1. bimalleolar fracture requiring fixation of any two malleoli (i.e. lateral/medial, medial/posterior, lateral/posterior)
   2. bimalleolar equivalent SER4 fractures (lateral malleolus fracture requiring fixation and no medial or posterior malleolus fixation)
   3. trimalleolar fracture with fixation of at least two malleoli (i.e. lateral/medial, medial/posterior, lateral/posterior)
3. Operative treatment of an isolated lower extremity unicondylar tibial plateau fracture (AO/OTA 41B1, Schatzker Type 1or 4) without joint impaction.

Exclusion Criteria:

1. Gustilo Type III injuries or soft tissue injury of either lower extremity that would contra-indicate immediate or delayed WB
2. Syndesmotic injuries/fixation
3. Osteoporosis as defined by treatment with a bisphosphonate and/or other osteoporosis medications, including Prolia and Forteo; or a prior fragility fracture (e.g., spine compression, proximal humerus, distal radius, femoral neck/intertrochanteric fracture)
4. Neuropathy, defined as diagnosis of peripheral neuropathy in medical record, neuropathic foot ulcer, or diminished or absent plantar sensation to light touch.
5. Pathologic fracture related to neoplasm
6. Fractures and dislocations to the ipsilateral or contralateral lower limb that prevent weight bearing as tolerated after fist post-op visit
7. Other contra-indication to immediate or delayed weight bearing (e.g., ipsilateral fracture effecting weight bearing status such as a calcaneus fracture); fractures of the ipsilateral lower extremity that would not affect WB status may be included (e.g., proximal femur, femoral shaft or tibia shaft fractures)
8. Any upper limb injury that would limit upper extremity weight bearing (e.g., surgical neck fracture of proximal humerus)
9. Injuries to other body systems that would affect the ability to comply with either WB protocol (e.g., spinal cord injury; severe TBI; major abdominal or chest injury)
10. Patient has third degree burns on >10% total surface area affecting the study limb
11. Tibial plateau fractures that are required to wear a locking brace or fractures that require fixed immobilization beyond four weeks (e.g., cast)
12. Non-ambulatory pre-injury
13. Pre-injury limitation to ROM of ipsilateral hip, knee or ankle
14. Morbidly obese (BMI ≥40)
15. Documented psychiatric disorder requiring admission in perioperative period
16. Severe problems with maintaining follow-up (e.g., patients who are prisoners or homeless at the time of injury or who are intellectually challenged without adequate family support)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of Study Related Complications Experienced | 12 months
  Re-admissions for a limb related issue and all re-operations on the study limb will be prospectively tracked by the Research Coordinators by routinely scanning hospital admission and orthopaedic surgery logs to identify all admissions and same day surgeries of patients actively enrolled in the study. Complications include loss of reduction and hardware failure, infection, non-union, malunion and fusion.
Return to Usual Major Activity and Work Productivity | 12 months
  Participants will be asked what they were doing most of the time during the previous two weeks (working/active duty, laid off/looking for work, going to school, taking care of a home, etc.). If participants are working, the Work Productivity and Activity Impairment (WPAI) questionnaire will be administered.The WPAI measures work time missed and work and activity impairment because of a specified health problem during the past 7 days (http://www.reillyassociates.net/WPAI_SHP.html).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reider, PhD, Principal Investigator — Major Extremity Trauma Research Consortium
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco Medical Center, San Francisco, California
  - Methodist Hospital, Indianapolis, Indiana
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Hennepin County Medical Center / Regions Hospita, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Washington/Harborview Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Data sharing beyond manuscripts and scientific presentations will be processed through the METRC website in the short term. Currently, a standard form will be available for researchers outside METRC to request access to final data generated from METRC studies. These requests will be transmitted to the METRC Coordinating Center for initial review to make sure the relevant materials are provided in support of the request. METRC is committed to making data as widely available as possible while safeguarding the privacy of study participants and protecting the intellectual property of the Consortium.
  Data will only be made available after it is completely stripped of identifiable information such as dates, geographic locators, and any other event information which is sufficiently rare as to make it possible to deduce the identity of an individual participant. When necessary for complete de-identification, data may be grouped.
Time Frame: Once study activities are complete.
Access Criteria: See plan description.